CLINICAL TRIAL: NCT03521713
Title: A Randomized, Active Comparator-Controlled, Parallel-Group, Single-Blind, Multicenter, Phase III Study to Evaluate the Efficacy, Safety and Immunogenicity of Subcutaneous Eporon Versus Epoetin Alfa (Eprex) in the Treatment of Anemia Associated With Chronic Renal Failure in Pre-dialysis Patients
Brief Title: To Evaluate the Efficacy, Safety, and Immunogenicity of Subcutaneous Eporon Versus Epoetin Alfa (Eprex)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAEPO_ANE_III
Record Dates: First submitted 2017-02-21; First posted 2018-05-11 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only investigators will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPORON (Experimental): <Part 1 Treatment Period> Week 1 to Week 24 Initial Phase (Week 1 to Week 4) : 50 IU/kg of Erythropoietin Alpha, three times a week (3 x 50 IU/kg/week) No dose adjustments will be permitted during the first 4 weeks of the study. Maintenance Phase (Week 5 to Week 24) The dose will be adjusted to maintain Hb levels between 10 and 12 g/dL.
  <Part 2 Treatment Period> : Week 25 to Week 52 The dose of Erythropoietin Alpha will be adjusted to maintain hemoglobin levels between 10 and 12 g/dL as subcutaneous administration in accordance with the given dosing algorithm. The further details are the same as those for maintenance phase of Part 1 Treatment Period.
  Interventions: Drug: EPORON
- EPREX (Active Comparator): <Part 1 Treatment Period> Week 1 to Week 24 Initial Phase (Week 1 to Week 4) : 50 IU/kg of Erythropoietin Alpha, three times a week (3 x 50 IU/kg/week) No dose adjustments will be permitted during the first 4 weeks of the study. Maintenance Phase (Week 5 to Week 24) The dose will be adjusted to maintain Hb levels between 10 and 12 g/dL.
  <Part 2 Treatment Period> : Week 25 to Week 52 The dose of Erythropoietin Alpha will be adjusted to maintain hemoglobin levels between 10 and 12 g/dL as subcutaneous administration in accordance with the given dosing algorithm. The further details are the same as those for maintenance phase of Part 1 Treatment Period.
  Interventions: Drug: EPREX

INTERVENTIONS:
Drug: EPORON — * Strength : 3000 IU/0.3 mL, 5000 IU/0.5 mL, 6000IU/0.6 mL
  * Formulation : Solution in PFS
  Other Names: Erythropoietin Alpha
  Arms: EPORON
Drug: EPREX — * Strength : 2000 IU/0.3 mL, 3000 IU/0.5 mL, 4000IU/0.6 mL
  * Formulation : Solution in PFS
  Other Names: Erythropoietin Alpha
  Arms: EPREX

SUMMARY:
This study is to evaluate 24-week efficacy and 52 week immunogenicity of subcutaneous Eporon versus Epoetin Alfa (Eprex) in the treatment of anemia associated with chronic renal failure in pre-dialysis patients. A total of 214 patients will be enrolled in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Glomerular Filtration Rate <60 mL/min/1.73m2 (estimated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)
* Hemoglobin (Hb) level in the range of ≥7 g/dL and <10 g/dL at screening
* Erythropoiesis Stimulating Agent (ESA) naïve subjects or previously treated subjects with ESA-free period of >3 months (in case of pre-treatment with long-acting ESA such as pegylated epoetin, the long-acting ESA-free period of >6 months)

Exclusion Criteria:

* Subjects who have received steady dialysis or subjects who are currently on dialysis
* Subjects who have rapid progression of chronic renal failure (as per investigators' discretion; e.g., a GFR decrease of >20% within 12 weeks prior to screening)
* Subjects who have already undergone renal transplantation or who are scheduled for renal transplantation

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Mean Absolute Change in Hb levels | Week -2~Week 1 (Prior to Dose), Week 1, Week 21, Week 22, Week 23, Week 24
  The primary endpoint is the mean absolute change in Hb levels between the screening/baseline period (Week -2 to Day 1 of Week 1) and the evaluation period (Week 21 to Week 24).
  Hb level at screening/baseline period is defined as the mean of the Hb measurements at screening and on Day 1 of Week 1 (prior to dosing). Hb level at evaluation period is defined as the mean of the Hb measurements at Week 21, 22, 23, and 24 (in detail, Day 1 of Week 21, Day 1 of Week 22, Day 1 of Week 23, and Day 1 of Week 24).

SECONDARY OUTCOMES:
Hemoglobin Responder Rate | Week -2~Week 1 (Prior to Dose), Week 1, Week 21, Week 22, Week 23, Week 24
Mean EPO dosage (Week 1 to Week 24) | Week 1 ~ Week 24
Mean EPO dosage (Week 21 to Week 24) | Week 21 ~ Week 24

OTHER OUTCOMES:
Safety: Any adverse events | Week 1 to Week 52
  Any adverse events
Immunogenicity: Anti-drug antibody (ADA) response by Week 52 compared to baseline (Week -2~Week 1 (Prior to Dose)) | (Week -2~Week 1 (Prior to Dose)), Week 52
  Anti-drug antibody (ADA) response by Week 52 compared to baseline (Week -2~Week 1 (Prior to Dose))

CONTACTS AND LOCATIONS:
Overall Officials: Turgay Arinsoy, MD, Study Chair — Gazi University Medical Faculty
Locations (1):
- Gazi University Medical Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No